CLINICAL TRIAL: NCT02652338
Title: Influence of a Specific Micronutrient Combination on Symptom Awareness and Heart Rhythm in Patients With Cardiac Arrhythmia
Brief Title: Dietary Supplement on Symptom Awareness and Heart Rhythm in Patients With Cardiac Arrhythmia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trommsdorff GmbH & Co. KG (Industry)
Collaborators: Bonn Education Association for Dietetics r.A., Cologne, Germany (Industry)
Responsible Party: Principal Investigator, Christine Metzner Prof. Dr. Dr., chief Executive Officer, Bonn Education Association for Dietetics r.A., Cologne, Germany, Trommsdorff GmbH & Co. KG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MNC-01
Record Dates: First submitted 2015-12-16; First posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Cardiac Arrhythmia
Keywords: heart rhythm disturbances and symptoms; dietary supplement
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MNC-01 (Active Comparator): potassium, magnesium, and vitamins (MNC-01)
  Interventions: Dietary Supplement: MNC-01
- Placebo (Placebo Comparator): cellulose, microcrystalline [NF], HPMC E15,
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MNC-01 — twice daily 2 tablets with appr. 200 ml still water or tap water; duration: 6 weeks
  Arms: MNC-01
Dietary Supplement: Placebo — twice daily 2 tablets with appr. 200 ml still water or tap water; duration: 6 weeks
  Arms: Placebo

SUMMARY:
The main aim of this study, which was carried out in two parallel groups, is testing the efficacy of a specific micronutrients combination in adults with heart rhythm disturbances and accompanying symptoms.

It is therefore the investigators hypothesis that daily oral administration of the specific micronutrients combination will lead to a decrease of symptoms awareness and to a reduction of heart rhythm disturbances in adults with or without structural heart disease. The principal endpoints will be a decrease in the total score of symptoms awareness.

ELIGIBILITY:
Inclusion Criteria:

* PVB in the long-term ECG recording (registration at least 18 hours): at least 500 PVB/24 h or Supraventricular tachycardia (≥10 episodes/24h, outside sporting activity) or SVPB with vegetative symptoms (increased sweating, inner unrest, shaky hands, red dermographism) and no cardial pretreatment

Exclusion Criteria:

* Left ventricular ejection fraction [EF] ≤ 40 %
* Therapy with spironolactone > 50 mg/d
* Therapy with torasemide > 20 mg/d
* Supplementation or therapy with dietary supplements or drugs which contain vitamins and minerals (above all potassium and magnesium)
* Creatinine in the serum [i. S.]:≥ 1,4 mg/dl (men), ≥ 1,2 mg/dl (women)
* Potassium i. S. ≤ 3,4 mmol/l and > 5,4 mmol/l
* Magnesium i. S. ≤ 0,7 mmol/l and > 1,0 mmol/l
* Acute and chronic diarrhea
* Hyperthyroidism anamnestic or due to the current TSH (thyroid stimulating hormone)-value
* Pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the changes in the perception of six symptoms | end week 3 and week 6
  at baseline, at follow-up visit 4 (at the end of week three) and at follow-up visit 5 (at the end of study) by visual analogue scale [VAS]: complete summary to a total score value in comparison to baseline

SECONDARY OUTCOMES:
symptom awareness and responder rate | end week 6
  the responder rates of the changes, measured by the amount of patients with a reduction of the total score value at follow-up visit 5 (at the end of study) in comparison to baseline of at least 20%
symptom awareness and changes during the study | end week 3 and week 6
  evaluation of the changes in the awareness of six symptoms, namely: irregular heartbeat, palpitations, heart stumbling, sweating, dyspnea, and anxiety or panic attacks at baseline, at follow-up visit 4 (at the end of week three) and at the end of week six by VAS and summary to a total score value
absolute reduction in premature ventricular beat (PVB) | end week 3 and 6 week
  the absolute reduction of the PVB in 24 hours at follow-up visit 4 (at the end of week three) and follow-up visit 5 (at the end of study) in comparison to baseline
relative reduction of the premature ventricular beat (PVB) | end week 3 and week 6
  the relative reduction of the PVB in 24 hours at follow-up visit 4 (at the end of week three) and follow-up visit 5 (at the end of study) in comparison to baseline
responder rate of the premature ventricular beat (PVB) | end week 3 and week 6
  the responder rate measured by the amount of patients with a reduction of the PVB of at least 5 % at the end of study
absolute reduction of supraventricular premature beats (SVPB) | end week 3 and week 6
  the absolute reduction of the SVPB in 24 hours in combination with a reduction of the awareness of the six symptoms
relative reduction of supraventricular premature beats (SVPB) | end week 3 and week 6
  the relative reduction of the SVPB in 24 hours in combination with a reduction of the awareness of the six symptoms
responder rate | end week 3 and week 6
  the responder rate, measured by the amount of patients with a reduction of the PVB of at least 5 % at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Christine Metzner, Prof. MD, Study Chair — Bonn Education Association for Dietetics r. A.
Locations (1):
- Elke Parsi assoc. Prof. MD, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Parsi E, Bitterlich N, Winkelmann A, Rosler D, Metzner C. Dietary intervention with a specific micronutrient combination for the treatment of patients with cardiac arrhythmias: the impact on insulin resistance and left ventricular function. BMC Cardiovasc Disord. 2018 Dec 3;18(1):220. doi: 10.1186/s12872-018-0954-6. PMID 30509185